CLINICAL TRIAL: NCT05088876
Title: Paracetamol in Addition to WHO Step III Opioids in Chronic Cancer Pain Control - a Randomized, Double-blind, Placebo-controlled, Non-inferiority Study
Brief Title: Paracetamol in Addition to WHO Step III Opioids in Chronic Cancer Pain Control
Acronym: ParOP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BASEC-ID: 2021-01518
Record Dates: First submitted 2021-10-05; First posted 2021-10-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Active Comparator)
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Blinded withdrawal of regular co-medication with paracetamol
  Arms: Placebo
Drug: Paracetamol — Paracetamol in the dose already used
  Arms: Paracetamol

SUMMARY:
Blinded withdrawal of regular co-medication with paracetamol in chronic pain patients under strong opioids on pain control.

DETAILED DESCRIPTION:
Chronic pain patients receiving a strong opioid in combination with paracetamol in a minimum dose of 1.5 g/day will be randomized to receive either paracetamol in the dose already prescribed (group "paracetamol") or an identically looking placebo (group "placebo") using the same schedule during the first study phase (days 1-7). In the second study phase (days 8-14) paracetamol or placebo will be stopped in both arms to assess the effect of pill withdrawal on pain control.

Next to baseline the patients will be instructed to use a pain diary to rate their pain during the study and also document the required opioid rescue doses. Further assessments will include adverse events, subjective ratings of quality of sleep, overall feeling of functioning and quality of life. At the screening visit, patients will also be asked to rate their expected changes in pain relief as a result of co-treatment with paracetamol. At the completion of the study, patients will be asked about their preference and whether, overall, they felt their pain was more poorly controlled during the study.

Adherence will be checked by pill count and measurement of paracetamol blood concentrations. Genotyping of OPRM1, COMT and relevant CYP enzymes and opioid blood concentrations will be assessed as co-variates for pain control.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients receiving a WHO step III opioid (i.e. morphine, oxycodone, methadone, fentanyl, hydromorphone, or buprenorphine) in combination with paracetamol (minimum dose 1.5 g/day)
* Age ≥ 18 at screening
* Ability to understand the study procedures and to provide written informed consent
* Stable analgesia before randomisation, defined as no required changes in the analgesic treatment during the previous 7 days

Exclusion Criteria:

* Participation in another interventional trial within 30 days prior to randomisation, with the exception of cancer treatment trials
* Changes of the dosage or start of other (co-)analgesics (e.g. tricyclic antidepressants, neuroleptics, nonsteroidal anti-inflammatory drugs (NSAIDs), dipyrone), within the last 7 days preceding randomisation
* Surgery within the 14 days preceding randomisation or surgery planned within the duration of the study
* Any circumstances, comorbidities or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
VAS score (average pain intensity) | Study day 7

SECONDARY OUTCOMES:
Average pain using the Brief Pain Inventory (BPI) | On each study day, up to 14 days
Minimum pain using the Brief Pain Inventory (BPI) | On each study day, up to 14 days
Worst pain using the Brief Pain Inventory (BPI) | On each study day, up to 14 days
Current pain using the Brief Pain Inventory (BPI) | On each study day, up to 14 days
Average pain using the Brief Pain Inventory (BPI) | During the last four days of each study phase (days 4-7 und 11-14)
Minimum pain using the Brief Pain Inventory (BPI) | During the last four days of each study phase(days 4-7 und 11-14)
Worst pain using the Brief Pain Inventory (BPI) | During the last four days of each study phase (days 4-7 und 11-14)
Current pain using the Brief Pain Inventory (BPI) | During the last four days of each study phase (days 4-7 und 11-14)
Cumulative dose of rescue medication used | On each study day, up to 14 days
Cumulative dose of rescue medication used | During the last four days of each study phase (days 4-7 und 11-14)
Number of rescue medication used | On each study day, up to 14 days
Number of rescue medication used | During the last four days of each study phase (days 4-7 und 11-14)
Percentage increase in pain compared to baseline | During each study phase (days 1-7 and days 8-14)
Percentage of patients meeting the predefined pain threshold | During each study phase (days 1-7 and days 8-14)
Subjective ratings of quality of sleep using the Brief Pain Inventory (BPI) | At baseline and during each study phase (days 1-7 and days 8-14)
Subjective ratings of quality of life using the EQ-5D-5L questionnaire | At baseline and during each study phase (days 1-7 and days 8-14)
Subjective ratings of functioning using the Brief Pain Inventory (BPI) and the EQ-5D-5L questionnaire | At baseline and during each study phase (days 1-7 and days 8-14)
Patients' expectation regarding pain relief from paracetamol prior to study treatment paracetamol using the Expectation for Treatment Scale (ETS) | Prior to study treatment
  Five-item ETS with each item rated on a 4-point scale ranging from 1 to 4 (partially disagree, partially agree, agree and definitely agree)
Question about participant's preference | At day 7 and 14
  Study vs. baseline
Participant's impression of change | At day 7 and 14
  11-point scale tool between -5 ="very much worse" and +5 ="completely recovered"
Participants' guess regarding their assigned group (verum or placebo) | At day 7 and 14
Assessment of serious adverse events | During each study phase (days 1-7 and days 8-14)
Assessment of specific adverse events: nausea/vomiting | During each study phase (days 1-7 and days 8-14)
Assessment of specific adverse events: drowsiness | During each study phase (days 1-7 and days 8-14)
Assessment of specific adverse events: appetite | During each study phase (days 1-7 and days 8-14)
Assessment of specific adverse events: constipation | During each study phase (days 1-7 and days 8-14)
Assessment of other adverse events | During each study phase (days 1-7 and days 8-14)
Number of withdrawals from study or treatment | During each study phase (days 1-7 and days 8-14)
Time (days) of stable pain control | During whole study (days 1-14)
Patients' potential to develop hepatotoxicity (investigation of risk factors) | During whole study (days 1-14)
% hours with pain/24h | On each study day, up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Liakoni, Principal Investigator — Inselspital, Bern University Hospital
Locations (2):
- Switzerland (2):
  - Kantonsspital Baden, Baden
  - Inselspital, Bern University Hospital, Bern

IPD SHARING:
Plan to Share IPD: Yes
Data that relates to individual, primary publications (and not the whole study database as such) will be deposited in the Bern Open Repository and Information System (BORIS). All efforts will be made to protect privacy and to de-identify the data. Data will be shared on request under the following conditions: A meaningful study question by the requester, outline of the planned analyses, valid methodology, signed data sharing agreement that contains a confidentiality agreement in case of sensitive data.
URL: https://boris.unibe.ch/

REFERENCES:
- [Derived] Kotoula C, Wertli MM, Streitberger K, Rothschild SI, Limacher A, Hammann F, Krahenbuhl S, Haschke M, Liakoni E. Efficacy of paracetamol added to WHO step III opioids in chronic pain control: study protocol for a randomised, double-blind, placebo-controlled, non-inferiority, multicentre study in Switzerland. BMJ Open. 2025 Dec 31;15(12):e107360. doi: 10.1136/bmjopen-2025-107360. PMID 41475826